CLINICAL TRIAL: NCT05123833
Title: The Optimal Urethral Coverage in Hypospadias Repair: Dartos Fascia Versus Tunica Vaginalis Flap? A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hypospadias-UC
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Pediatric Disorder; Hypospadias; Congenital Hypospadia; Urologic Diseases
Keywords: Hypospadias repair; Tunica Vaginalis Flap; Dartos Fascia; Fistula
MeSH Terms: conditions — Hypospadias; Urologic Diseases; Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dartos Fascia (Active Comparator): Dartos flap is used as a covering layer for urethra during repair of hypospadias
  Interventions: Procedure: Hypospadias repair
- Tunica Vaginalis (Active Comparator): Tunica Vaginalis Flap is used as a covering layer for urethra during repair of hypospadias
  Interventions: Procedure: Hypospadias repair

INTERVENTIONS:
Procedure: Hypospadias repair — surgical repair of hypospadias

SUMMARY:
To explore the optimal urethral coverage in hypospadias repair by comparing the success rate of both covering techniques: Dartos fascia versus Tunica Vaginalis flap.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 months.
* Distal, mid-shaft penile hypospadias.

Exclusion Criteria:

* Glanular hypospadias.
* Penoscrotal, Scrotal & Perineal hypospadias.
* Recurrent cases.

Ages: 6 Months to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — males less than 12 years
Enrollment: 88 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Fistula | Within the first three months after surgery.
  Fistula prevalence will be recorded as a complication after surgery

SECONDARY OUTCOMES:
Cosmetic outcome | Within the first three months after surgery.
  Patients' parents reported cosmetic outcomes will be evaluated using The Pediatric Penile Perception Score (PPPS).

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No